CLINICAL TRIAL: NCT06998407
Title: A Phase 1/2, First-in-human Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Antitumor Activity of AVZO-023 as a Single Agent, and in Combination With AVZO-021 and/or Endocrine Therapy in Patients With Advanced Solid Tumors
Brief Title: Study of AVZO-023 as a Single Agent and in Combination With AVZO-021, and/or Endocrine Therapy in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Avenzo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AVZO-023-1001
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: HR+/HER2- Breast Cancer; HR+, HER2-, Advanced Breast Cancer
MeSH Terms: interventions — Fulvestrant; Letrozole

STUDY DESIGN:
Intervention Model Description: Phase 1 dose-escalation Phase 2 dose-expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1, monotherapy (Part 1A) and food effect (Experimental): Escalating doses of twice daily, oral AVZO-023 in 28-day cycles, with addition of fulvestrant
  Interventions: Drug: Fulvestrant; Drug: AVZO-023
- Phase 1, combination (Parts 1B) (Experimental): Escalating doses of twice daily, oral AVZO-023 in combination with once daily, oral AVZO-021 in 28-day cycles, with addition of fulvestrant
  Interventions: Drug: AVZO-021; Drug: Fulvestrant; Drug: AVZO-023
- Phase 1, combination (Parts 1C) (Experimental): Escalating doses of twice daily, oral AVZO-023 in combination with once daily, oral AVZO-021, with once daily, oral letrozole in 28-day cycles
  Interventions: Drug: AVZO-021; Drug: Letrozole; Drug: AVZO-023
- Phase 2, combination (Cohorts 2A, 2B, 2C, and 2D) (Experimental): Oral doses of AVZO-023 in 28-day cycles at the RP2D determined in Part 1B/1C, in combination with:
  2A) letrozole
  2B) fulvestrant
  2C) AVZO-021 plus fulvestrant
  2D) AVZO-021 plus letrozole
  Interventions: Drug: AVZO-021; Drug: Fulvestrant; Drug: Letrozole; Drug: AVZO-023

INTERVENTIONS:
Drug: AVZO-021 — AVZO-021 is an oral selective CDK2 inhibitor
  Arms: Phase 1, combination (Parts 1B); Phase 1, combination (Parts 1C); Phase 2, combination (Cohorts 2A, 2B, 2C, and 2D)
Drug: Fulvestrant — Antineoplastic agent, estrogen receptor antagonist
  Other Names: Faslodex
  Arms: Phase 1, combination (Parts 1B); Phase 1, monotherapy (Part 1A) and food effect; Phase 2, combination (Cohorts 2A, 2B, 2C, and 2D)
Drug: Letrozole — Antineoplastic agent, aromatase inhibitor
  Other Names: Femara
  Arms: Phase 1, combination (Parts 1C); Phase 2, combination (Cohorts 2A, 2B, 2C, and 2D)
Drug: AVZO-023 — AVZO-023 is an oral selective CDK4 inhibitor

SUMMARY:
This study, the first clinical trial of AVZO-023, aims to determine the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, maximum tolerated dose, and anti-tumor effects of AVZO-023 in patients with advanced solid tumors. AVZO-023 is an oral medication that inhibits cyclin-dependent kinase 4 (CDK4).

DETAILED DESCRIPTION:
AVZO-023 is an oral, potent, and selective inhibitor of CDK4. AVZO-021 is an oral, potent, and selective inhibitor of CDK2 that is currently being investigated in a global Phase 1/2 study in patients with advanced hormone receptive positive (HR+)/human epidermal growth factor receptor 2 negative (HER2-) breast cancer (NCT05867251).

In Phase 1, the safety and tolerability of AVZO-023 in patients with HR+/HER2- locally advanced or metastatic breast cancer (mBC) will be assessed. The goal of Phase 1 is to determine the MTD/preliminary RP2D of AVZO-023 for use as monotherapy and in combination with AVZO-021 with or without endocrine therapy (ET).

Phase 2 will assess the antitumor activity and confirm the RP2D of AVZO-023 in combination therapy in patients with HR+/HER2- locally advanced or mBC.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female aged ≥ 18 years old at screening with Eastern Cooperative Oncology Group (ECOG) 0-1 and life expectancy > 3 months
* Patients with histologically or cytologically proven advanced malignancies of preferred indications
* Measurable disease (as assessed by investigator using RECIST v1.1) is preferred in Phase 1 dose escalation, unless otherwise specified in the protocol, and in all patients in Phase 2. Bone only disease is allowed in dose escalation.
* Agree to provide molecular test report results to confirm eligibility and archival tumor samples and/or fresh biopsy, as applicable
* Adequate renal, liver, and bone marrow function

Key Exclusion Criteria:

* Patients should not have received any prior selective investigational CDK (CDK2, CDK4, CDK2/4, CDK2/4/6) inhibitors
* Has known active brain metastasis (have either previously untreated intracranial CNS metastasis or previously treated intracranial central nervous system (CNS) metastasis with radiologically documented new or progressing CNS lesions) or leptomeningeal disease
* Other concurrent invasive malignancy or a prior invasive malignancy for which treatment was completed within 3 years before the first dose on study except for adequately treated basal cell or squamous cell skin cancer, carcinoma in situ, or colorectal adenomatous polyps
* Last anticancer treatment within 2 weeks (4 weeks for biologic, immunotherapy or ADC) or 5 half-lives of the drug, whichever is shorter, prior to first dose on study
* Major surgery within 4 weeks prior to first dose on study
* Have received radiotherapy with a limited field of radiation for palliation within 7 days of the first dose of study treatment, except for patients receiving whole brain radiotherapy, which must be completed at least 4 weeks prior to the first dose of study treatment. Patients must have recovered from all radiation-related toxicities, not require corticosteroids, and not have active radiation pneumonitis
* Strong or moderate CYP3A4 inhibitors or inducers within 2 weeks or 5 half-lives of the drug, whichever is shorter, prior to first dose on study
* History of serious cardiovascular conditions within 6 months prior to first dose on study
* Unresolved toxicities from prior therapy greater than Grade 1 (per CTCAE version 5.0) (with exceptions of alopecia, vitiligo, and ≤ Grade 2 peripheral neuropathy) prior to the first dose on study
* History of drug-induced pneumonitis/interstitial lung disease
* Confirmed loss of function mutation or deletion of Rb1 gene

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Dose Limiting Toxicities (DLTs) during the first cycle (Phase 1) | Cycle 1 (28 Days)
  Number of participants with DLTs assessed for severity using CTCAE v5.0 criteria will be summarized by dose level.
Number of Participants with Treatment Emergent Adverse Events (TEAEs) and lab abnormalities (Phase 1) | From baseline until end of study treatment or study completion (approximately 2 years)
Determine the Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) (Phase 1) | Approximately 16 months
Objective Response Rate (ORR) (Phase 2) | From baseline through disease progression or study completion (approximately 2 years)
  Defined as the proportion of patients with a confirmed Complete Response (CR) or Partial Response (PR), as determined by the investigator by radiographic disease assessment according to RECIST v1.1.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) (Phase 1) | From baseline through disease progression or study completion (approximately 2 years)
Duration of response (DOR) (Phase 1 and Phase 2) | From baseline through time to event on study or study completion (approximately 2 years)
  Defined as the time from the first confirmed response to radiologic/objective progression.
Progression Free Survival (PFS) (Phase 1 and Phase 2) | From baseline through time to event on study or study completion (approximately 2 years)
  Defined as the time from study drug treatment to death or disease progression, as determined by the investigator by radiographic disease assessment according to RECIST v1.1.
Overall Survival (OS) (Phase 1 and Phase 2) | Approximately 76 months
  Defined as the time from study drug treatment initiation to death from any cause.
Disease control rate (DCR) (Phase 1 and Phase 2) | From baseline through disease progression or study completion (approximately 2 years)
  Defined as the proportion of patients who achieve tumor relief (CR or PR) and stable disease (SD) after treatment; calculated as the sum of CR, PR, and SD.
Clinical benefit rate (CBR) (Phase 1 and Phase 2) | From baseline through disease progression or study completion (approximately 2 years)
  Defined as the percentage of advanced cancer patients who achieve CR, PR, or at least six months of SD after treatment.
PK Parameters: Maximum plasma concentration (Cmax) (Phase 1) | Day 1 and Day 15 of Cycle 1 (each cycle is 28 days)
PK Parameters: Time to maximum plasma concentration (Tmax) (Phase 1) | Day 1 and Day 15 of Cycle 1 (each cycle is 28 days)
PK Parameters: Elimination half-life (t1/2) (Phase 1) | Day 1 and Day 15 of Cycle 1 (each cycle is 28 days)
PK Parameters: Area under the plasma concentration-time curve from time 0 to last measurable concentration (AUC 0-last) (Phase 1) | Day 1 and Day 15 of Cycle 1 (each cycle is 28 days)
Determination of RP2D (Phase 2) | Approximately 16 months
Number of Participants with Treatment Emergent Adverse Events (TEAEs) and lab abnormalities (Phase 2) | From baseline until end of study treatment or study completion (approximately 2 years)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Avenzo Therapeutics Recruiting Site, Los Angeles, California
  - Avenzo Therapeutics Recruiting Site, New Haven, Connecticut
  - Avenzo Therapeutics Recruiting Site, Boston, Massachusetts
  - Avenzo Therapeutics Recruiting Site, New York, New York
  - Avenzo Therapeutics Recruiting Site, Cleveland, Ohio
  - Avenzo Therapeutics Recruiting Site, Nashville, Tennessee
  - Avenzo Therapeutics Recruiting Site, Houston, Texas
  - Avenzo Therapeutics Recruiting Site, San Antonio, Texas
  - Avenzo Therapeutics Recruiting Site, Fairfax, Virginia